CLINICAL TRIAL: NCT07254611
Title: Combinazione HMA e Venetoclax Con Posaconazolo in Pazienti Affetti da Leucemia Acuta Mieloide: Studio Delle Concentrazioni Plasmatiche
Brief Title: Combination of HMA and Venetoclax With Posaconazole in Patients With Acute Myeloid Leukemia: A Study of Plasma Concentrations
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Patrizia Zappasodi, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: Prj_Venetoclax
Record Dates: First submitted 2025-11-17; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-08

CONDITIONS: AML (Acute Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Acute Myeloid Leukemia requires intensive chemotherapy treatment, usually followed by an allogeneic bone marrow transplant to reduce the risk of relapse. However, in elderly patients, intensive treatment is often not a feasible option due to the high toxicity, which limits its use. Recently, a combination of hypomethylating agents (HMAs, 5-azacitidine or decitabine), which have a low toxicity profile, and venetoclax, a potent inhibitor of the anti-apoptotic protein Bcl2, has been approved for patients with Acute Myeloid Leukemia who are not candidates for intensive therapy. This combination has shown a significant survival advantage compared to the use of HMA alone (Di Nardo, NEJM 2020). Even in the difficult setting of relapsed/refractory patients, the combination of venetoclax with an HMA agent has led to high rates of global response and good-quality response (global responses 64%, of which 50% were complete responses or with incomplete hematopoietic recovery), as well as disease-free survival rates of 8.9 months for responsive patients, offering many the option for allogeneic transplantation (Aldoss, Haematologica 2018).

However, the venetoclax-HMA combination is associated with hematological toxicity, characterized by deep and prolonged cytopenias, particularly in non-responsive diseases but also after achieving complete remission. Therefore, the risk of infection during periods of severe neutropenia is high. For this reason, although the need for infection prophylaxis in this therapeutic regimen is not yet well defined, it is common practice to administer antifungal prophylaxis with posaconazole, at least during the first two months of therapy or until neutropenia resolves. Posaconazole has been shown to reduce fungal complications during treatment for active Acute Leukemia stages. An increased incidence of invasive fungal infections has been reported in patients with active disease (refractory or at diagnosis). However, this choice must take into account the pharmacological interactions with venetoclax, as posaconazole is a strong inhibitor of cytochrome P3A4 activity and may reduce venetoclax metabolism, thus increasing its plasma levels. To avoid excessive toxicity from venetoclax, its dosage must be adjusted.

Pharmacokinetic studies have shown that during prophylaxis therapy with posaconazole, treatment with venetoclax at doses of 50 or 100 mg was well tolerated. Therefore, based on the increased plasma levels of venetoclax, it is recommended that its dosage be reduced by at least 75% compared to the full dose (Agarwal, Clin Ther 2017).

The available pharmacokinetic studies evaluating venetoclax plasma levels in combination with posaconazole only consider levels after venetoclax has reached steady state (Agarwal, Clin Ther 2017). However, it is known that co-administration can alter venetoclax concentrations until a stable plasma level of posaconazole is reached. During this period, it is important to monitor venetoclax levels closely in order to adjust the dosage and avoid excessive exposure to the drug, thus reducing the risk of increased toxicity, but without excessively lowering plasma levels, which could compromise the treatment's efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with Acute Myeloid Leukemia undergoing standard treatment with the first cycle of the combination of Azacitidine or Decitabine and Venetoclax at the Hematology Clinic of the Fondazione IRCCS Policlinico San Matteo in Pavia.

Exclusion Criteria:

-

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients with Acute Myeloid Leukemia undergoing standard treatment with the first cycle of the combination of Azacitidine or Decitabine and Venetoclax at the Hematology Clinic of the Fondazione IRCCS Policlinico San Matteo in Pavia.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
To evaluate the proportion of patients who reach steady state on day 12. A blood sample will be collected before the administration of the first daily dose. | 12 DAYS
  To evaluate the proportion of patients who reach steady state on day 12. A blood sample will be collected before the administration of the first daily dose.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Lombardy, Italy